CLINICAL TRIAL: NCT05976932
Title: The Utility of Circulating Tumor DNA in Monitoring the Response to Pegylated Liposomal Doxorubicin in Platinum-resistant Ovarian Cancer
Brief Title: Circulating Tumor DNA Monitoring in Platinum-resistant Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaohua Wu, Director,Clinical Professor, Fudan University
Other Study IDs: 2210263-1
Record Dates: First submitted 2023-06-30; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Ovarian Cancer
Keywords: ctDNA; pegylated liposomal doxorubicin; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — liposomal doxorubicin; 1-dodecylpyridoxal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- treatment group: After enrollment, patients will receive standard treatment (pegylated liposomal doxorubicin) and follow-up strategy. Peripheral blood samples will be collected from all patients before treatment and 3 weeks after the first cycle of treatment，If necessary, Peripheral blood samples also be collected after 2 cycles of treatment.
  Interventions: Drug: pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin — All eligible subjects will receive the standard chemotherapy of pegylated liposomal doxorubicin monotherapy.
  Other Names: PLD

SUMMARY:
This observational study is conducted to assess the utility of circulating tumor DNA in monitoring the response to pegylated liposomal doxorubicin in platinum-resistant ovarian cancer，and evaluate the consistency of circulating tumor DNA with imaging and CA125 in platinum-resistant ovarian cancer.

DETAILED DESCRIPTION:
The goal of this study is to assess the utility of circulating tumor DNA in monitoring the response to pegylated liposomal doxorubicin in platinum-resistant ovarian cancer.This is a single-arm, single-center prospective clinical study.

After enrollment, patients will receive standard treatment (pegylated liposomal doxorubicin)and follow-up strategy. Peripheral blood samples will be collected from all patients before treatment and 3 weeks after the first cycle of treatment，If necessary, Peripheral blood samples also be collected after 2 cycles of treatment.Peripheral blood ctDNA will be tested for genetic variation based on next-generation sequencing (NGS).

Finally, this study will to evaluate the consistency of circulating tumor DNA with imaging and CA125 in platinum-resistant ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female, over 18 years of age;
2. Patients with histopathological diagnosis of high-grade serous epithelial ovarian cancer;
3. pathological report:phenotype of p53 mutation；or previous genetic tests of tumor tissue indicated TP53 gene mutations;
4. ECOG≤ 2;
5. Expected survival time ≥3 months;
6. The subjects were able to understand the study process and voluntarily joined the study.

Exclusion Criteria:

1. Pregnant and lactating patients;
2. Patients with severe or uncontrolled infections;
3. Patients who are allergic or intolerant to the investigational drug;
4. Patients who are enrolled in or within a month of another clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: platinum-resistant ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
the consistency of circulating tumor DNA with CT scan | at the beginning of Cycle 1 and 3 weeks after Cycle 1. If necessary, also including 3 weeks after Cycle 2（each cycle is 28 days）
  measuring the mutations of TP53，reporting the changes from baseline to 3 weeks after the first cycle, contrasting with CT scan changes，calculating Kappa value，and conducting a intrarater reliability

IPD SHARING:
Plan to Share IPD: No